CLINICAL TRIAL: NCT05039749
Title: Human Centric Lighting to Improve Patient Sleep Parameters: A Feasibility Study
Brief Title: Human Centric Lighting to Improve Patient Sleep Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landstuhl Regional Medical Center (U.S. Federal Agency)
Collaborators: TriService Nursing Research Program (Other)
Responsible Party: Principal Investigator, LTC Pauline Swiger, On-Site Principal Investigator, Landstuhl Regional Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LRMC CY16-36
Record Dates: First submitted 2021-06-25; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Central Lighting (HCL) Room (Experimental): This inpatient room was outfitted with lights that mimic the day/night cycle, thereby supporting circadian rhythm. Day time lights were automatically on during 0600 to 1900 and in use any time the patients would normally utilize their lights, with a goal of three hours of light exposure per day. The lights automatically transitioned to warmer toned evening lighting at 1900.
  Interventions: Device: Human Centric Lights
- Standard Hospital Lighting (SL) Room (No Intervention): The lighting in this room was standard florescent hospital lighting. The only changes in the lighting was the on/off settings normally associated with lighting.

INTERVENTIONS:
Device: Human Centric Lights — Bright light is emitted during the day from 06:00, then auto-dimmed light is used at night, beginning 19:00.
  Arms: Human Central Lighting (HCL) Room

SUMMARY:
Human centric lighting (HCL) is a technology that supports the body's circadian rhythm, as it can stimulate the sleep triggering hormone, melatonin, to improve sleep hygiene over standard lighting (SL), and promote recuperative sleep for a timely return-to-duty. In intensive care units, exposure to HCL has improved sleep measures. However, the effect in the medical surgical (MS) environment is unknown. The purpose of this study is to assess the feasibility of study procedures in MS setting and conduct a preliminary evaluation of the effect of light on inpatient sleep. Recruitment started November 2020 through April 2021. Data analysis is pending.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is an active duty service member, GS Civilian, Dependent or Retiree affiliated with the Army, Air Force or Navy.
* Patient who is informed by provider or anticipates being admitted for at least two nights.
* Patient who can read and speak English fluently (since surveys are not translated in any other language).

Exclusion Criteria:

* Patient with visual impairment which cannot be corrected with glasses or contact lenses such as complete blindness, (defined as inability to see light), or partial blindness (defined as very limited vision) such as patients with history of cataracts.
* Patient taking an oral medication for sleep.
* Patient receiving radioactive ionization treatment.
* Patient who requires isolation or palliative care.
* Patient recovering from head/neck or oral maxillofacial surgery that would impede saliva sample collection (i.e. jaw wiring, extensive gauze packing in oral cavity)
* Patient who reports status as a Department of Defense Contractor at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | During participant's inpatient stay, not to exceed 5 days.
  Assess the feasibility of measuring total sleep time in MS setting, using an actigraphy device.
Sleep Efficiency | During participant's inpatient stay, not to exceed 5 days.
  Assess the feasibility of measuring sleep efficiency in MS setting, using an actigraphy device.
Sleep Patterns | During participant's inpatient stay, not to exceed 5 days.
  Assess the feasibility of assessing sleep patterns in MS setting, using a Consensus Sleep Diary (CSD).
Dim Light Melatonin Onset - collection | During participant's inpatient stay, not to exceed 5 days.
  Assess the feasibility of collecting samples to assess dim light melatonin onset in MS setting, using passive drool saliva sampling.
Patient experience | One time - approximately a 5 to 15 minute interview
  Describe the patient's experience of participating in the study, in a MS setting, using a semi-structured interview (SSI).

SECONDARY OUTCOMES:
Dim Light Melatonin Onset - analysis | Collected during participant's inpatient stay, not to exceed 5 days.
  Conduct a preliminary evaluation of the effect of light on inpatient sleep using dim light melatonin onset saliva sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline A Swiger, PhD, Principal Investigator — US Army Landstuhl Regional Medical Ceneter
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT05039749/ICF_000.pdf